CLINICAL TRIAL: NCT06636695
Title: Clinical Efficacy of Platelet-Rich Plasma and Hyaluronic Acid Versus Hyaluronic Acid for Knee Osteoarthritis with MRI Analysis: a Randomized Controlled Trial
Brief Title: Clinical Efficacy of Platelet-Rich Plasma and Hyaluronic Acid Versus Hyaluronic Acid for Knee Osteoarthritis with MRI Analysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-2035
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP and HA (Experimental): Cellular-Matrix
  Interventions: Device: Cellular Matrix
- HA (Active Comparator): Orthovisc
  Interventions: Device: Orthovisc

INTERVENTIONS:
Device: Cellular Matrix — Group 1 (Cellular Matrix): Patients randomized to this group will be treated with two intra-articular injections of Cellular Matrix at D0 and M1.
  Arms: PRP and HA
Device: Orthovisc — Group 2 (HA): Patients randomized to this group will be treated with two intra-articular injections of HA alone provided by ORTHOVISC at D0 and M1
  Arms: HA

SUMMARY:
The study hypothesizes that the combination of Cellular Matrix PRP-HA is superior to Hyaluronic Acid (HA) alone, specifically from the Orthovisc Kit, in relieving pain and function associated with knee osteoarthritis.

The primary objective is to assess pain reduction following treatment. The secondary objectives, includes assessing the treatment's impact on function, stiffness, and overall quality of life for patients. In addition, non-invasive MRI will be employed at baseline and 12 months to evaluate changes in bone marrow edema, cartilage structure, and joint effusion. The study also aims to compare the safety of Cellular Matrix PRP-HA and HA.

ELIGIBILITY:
Inclusion Criteria:

* Participants fulfilling all of the inclusion criteria, listed below, are eligible to participate in this study:
* Patients between 40 and 80 years (inclusive) of age
* Femoro-tibial knee osteoarthritis defined
* OA grade 2-3 according to the Kellgren & Lawrence grading scale, as defined on knee radiographs (less than 6 months old: Antero-posterior view; lateral view and skyline view)
* Symptomatic knee osteoarthritis of a unilateral knee, characterized by pain at walking VAS ≥40 on a 0 to 100mm scale

  *Bilateral knee osteoarthritis is allowed, provided the contralateral knee is characterized by a maximum pain at walkingof 30 on a 0 to 100 mm scale and doesn't require systemic analgesic treatment, with the exception of paracetamol up to the maximum dose of 4 g per day
* Outpatient capableof walking 50 meters without assistance
* Signature of the informed consent form
* Capable of understanding the study's imperatives, as well as written instructions

Exclusion Criteria:

* Grade < 2 or > 3 OA according to the Kellgren & Lawrence gradingscale
* Viscosupplementation in the treatment site within the past 3 months
* Patients suffering from femoropatellar osteoarthritis
* Use of NSAIDs within the past 7 days
* Corticosteroid injection in the treatment site within the past 3 months
* Chronic use of corticosteroids (except those that are inhaled) or level III analgesics in the past 3 months and NSAID during the past month2 weeks
* PRP or PRP/HA injection in the past 12 months
* Any surgery of the knee planned within the next 12 months
* Unstable knee injury
* Systemic use of level III analgesics in the past 3 months
* History of allergy to HA
* Rheumatological disorders(exceptKOA)
* Clinical evidence of local inflammation such as redness or heat of the joint
* Current or medical history of autoimmunediseases
* Surgery or arthroscopy surgery in the affected knee within the past 3 months
* Local infection in the affected knee
* Haematologic or clotting disorders (thrombocytopenia platelet count <150,000 platelets/µ) or blood coagulation (deficit-blood dyscrasia)
* Anaemia (Haemoglobin <10g/dl)
* Anticoagulant treatment or Antiaggregant treatment
* Acute infection
* Immunosuppressive states
* Malignant disease
* Recent fever (within previous 2 weeks) or serious disorders (liver disease, active gastroduodenal ulcer, digestive haemorrhage, etc.)
* Pregnancy or breastfeeding or planning to become pregnant during the course of the study
* Uncontrolled diabeted
* Participation ongoing or in the past 3 months in another clinical trial
* Participation in another OA clinical study in the past year
* Refusal to sign or inability to give Informed Consent Inability to understand or comply with the requirements of the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Pain score | Baseline, Month 1, Month 2, Month 6, Month 12
  Visual Analogue Score (VAS) on a scale of 0 to 10. 10 being the worst possible pain.

SECONDARY OUTCOMES:
Quality of life | Baseline, Month 1, Month 2, Month 6, Month 12
  EQ-5D-5L. It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity: 1- no problem; 5- extreme problem
MRI | Baseline and Month 12
  Whole-Organ Magnetic Resonance Imaging Score (WORMS). WORMS evaluates 14 specific features. Each feature is scored on a scale: 0 = Normal; 1-6 = Increasing severity of abnormalities.
Function Score | Baseline, Month 1, Month 2, Month 6, Month 12
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The total WOMAC score is calculated by summing the scores from all three subscales: Pain, Stiffness, Physical Function. This can range from a minimum of 0 (indicating no symptoms) to a maximum of 96 (indicating severe symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Data available upon publication
Access Criteria: Request to lead author

REFERENCES:
- [Background] Campbell KA, Saltzman BM, Mascarenhas R, Khair MM, Verma NN, Bach BR Jr, Cole BJ. Does Intra-articular Platelet-Rich Plasma Injection Provide Clinically Superior Outcomes Compared With Other Therapies in the Treatment of Knee Osteoarthritis? A Systematic Review of Overlapping Meta-analyses. Arthroscopy. 2015 Nov;31(11):2213-21. doi: 10.1016/j.arthro.2015.03.041. Epub 2015 May 29. PMID 26033459
- [Background] Abate M, Verna S, Schiavone C, Di Gregorio P, Salini V. Efficacy and safety profile of a compound composed of platelet-rich plasma and hyaluronic acid in the treatment for knee osteoarthritis (preliminary results). Eur J Orthop Surg Traumatol. 2015 Dec;25(8):1321-6. doi: 10.1007/s00590-015-1693-3. Epub 2015 Sep 24. PMID 26403468
- [Background] Barac, B., N. Damjanov, and A. Zekovic, The new treatment approach in knee osteoarthritis: Efficacy of cellular matrix combination of platelet rich plasma with hyaluronic acid versus two different types of hyaluronic acid (HA). Int. J. Clin. Rheumatol., 2018. 13(5): p. 289-295.
- [Background] Pham T, van der Heijde D, Altman RD, Anderson JJ, Bellamy N, Hochberg M, Simon L, Strand V, Woodworth T, Dougados M. OMERACT-OARSI initiative: Osteoarthritis Research Society International set of responder criteria for osteoarthritis clinical trials revisited. Osteoarthritis Cartilage. 2004 May;12(5):389-99. doi: 10.1016/j.joca.2004.02.001. PMID 15094138
- [Background] Renevier, J.L., et al., "Cellular matrix™ PRP-HA": A new treatment option with platelet-rich plasma and hyaluronic acid for patients with osteoarthritis having had an unsatisfactory clinical response to hyaluronic acid alone: Results of a pilot, multicenter French study with long-term follow-up. Int. J. Clin. Rheumatol., 2018. 13(4): p. 230-238.
- [Background] LaBaze, D. and H. Li, Platelet Rich Plasma: Biology and Clinical Usage in Orthopedics, in Orthopedic Biomaterials : Progress in Biology, Manufacturing, and Industry Perspectives, B. Li and T. Webster, Editors. 2018, Springer International Publishing: Cham. p. 243-286.
- [Background] Yu W, Xu P, Huang G, Liu L. Clinical therapy of hyaluronic acid combined with platelet-rich plasma for the treatment of knee osteoarthritis. Exp Ther Med. 2018 Sep;16(3):2119-2125. doi: 10.3892/etm.2018.6412. Epub 2018 Jul 6. PMID 30186448